CLINICAL TRIAL: NCT05511272
Title: The Circadian Variability of Serum Progesterone During the Day of a Frozen Embryo Transfer in an Artificially Prepared Cycle and in a Modified Natural Cycle
Brief Title: The Circadian Variability of Serum Progesterone During the Day of a Frozen Embryo Transfer
Acronym: CIRCAPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1432022000124
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2022-07

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frozen embryo transfer cycle (Experimental): Patients who will undergo a frozen embryo transfer in the modified natural cycle and in an artificially prepared cycle will be included
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — four blood samples will be withdrawn from the participants during the day of their frozen embryo transfer cycle

SUMMARY:
Serum progesterone levels will be evaluated at four different time points during the day of an artificially prepared frozen embryo transfer cycle (HRT FET cycle) and a modified natural cycle frozen embryo transfer cycle (mNC FET cycle) (at 08:00, 12:00, 16:00 and 20:00).The pairwise percentage differences in serum progesterone levels for each patient will be calculated. The intra-day variability of progesterone will be analyzed using mixed models. Pregnancy outcomes will also be assessed. The sample size calculated consisted of 22 patients for the HRT-FET study and 22 patients for the mNC FET study.

DETAILED DESCRIPTION:
In the HRT FET, estradiol valerate (Progynova) will be administered for endometrial preparation. If the endometrial thickness will be ≥ 6,5 mm during an ultrasound scan planned following an initial period of estrogen priming, micronized vaginal progesterone will be started (Utrogestan 800 mg/d). The transfer of a single blastocyst will be performed on the 6th day of progesterone administration. In a modified NC FET, there is no intake of medication but endocrine and ultrasound monitoring during the proliferative phase. Ovulation trigger with hCG will be considered when a dominant follicle between 16 and 20 mm will be observed and when the endometrial thickness will be ≥ 6,5 mm. The transfer of a single blastocyst will take place on the 7th day after hCG injection.

Serum progesterone levels will be evaluated at four different time points during the day of an artificially prepared frozen embryo transfer cycle (HRT FET cycle) and a modified natural cycle frozen embryo transfer cycle (mNC FET cycle) (at 08:00, 12:00, 16:00 and 20:00). Pairwise percentage differences in serum progesterone levels for each patient will be calculated. The intra-day variability of progesterone will be analyzed using mixed models. Pregnancy outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 40 years old
* BMI ≥ 18.5 and ≤ 25,9 kg/m2
* The patient will undergo a hormone replacement therapy frozen embryo transfer cycle (HRT FET) or a modified natural cycle frozen embryo transfer cycle (mNC FET) according to the standard clinical practice in Brussels IVF
* In the HRT FET cycle the patient will be administered estradiol valerate and 6 days of micronized vaginal progesterone before the embryo transfer
* Adequate endometrial pattern (triple layer) and thickness (>6.5 mm) at the moment of planning of the transfer
* Single blastocyst embryo transfer
* Signed informed consent
* Non-smokers

Exclusion Criteria:

* Age > 40 (women > 40 years old demonstrated an enhanced rate of absorption of progesterone using vaginal tablets compared to younger patients)
* BMI ≥ 26 (serum progesterone levels on the day of embryo transfer are lower in overweight and obese women compared to those with normal weight)
* Patients who need to take vaginal estradiol valerate during the HRT FET cycle
* Intake of any experimental drug or any participation in any other clinical trial within 30 days prior to study start
* Mental disability or any other lack of fitness, in the investigator's opinion, to preclude subjects in or to complete the study.
* Current or recent substance abuse, including alcohol and tobacco (patients who stopped tobacco usage at least 3 months prior to screening visit would be allowed)
* Refusal or inability to comply with the requirements of the study protocol for any reason, including scheduled clinic visits and laboratory tests.
* Embryo transfer after IVM cycle, PGT or oocyte acceptance
* Uterine pathologies (fibroids, polyps, chronic endometritis), uterine malformations (septum, Mullerian malformation) and hydrosalpinx

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The existence of circadian variability of serum progesterone during the day of a frozen embryo transfer | the day of the embryo transfer (from 8 am to 8 pm)
  To evaluate if there is significant variability in circadian level of serum progesterone on the day of an artificially prepared frozen embryo transfer cycle and during the day of a modified natural frozen embryo transfer cycle

SECONDARY OUTCOMES:
Pregnancy outcomes after the frozen embryo transfer | from the day of the embryo transfer to 12 weeks of pregnancy
  To evaluate the Clinical pregnancy rate (CPR) in patients who underwent HRT FET or mNC FET. CPR is defined as a pregnancy documented by ultrasound at 6-8 gestational weeks that showed a gestational sac in the uterus
The critical progesterone threshold to optimize pregnancy outcomes | from the day of the embryo transfer to 12 weeks of pregnancy
  To evaluate the critical threshold of serum progesterone on the day of the FET below which pregnancy rates are significantly lower
The assessment of serum progesterone on the day of frozen embryo transfer | the day of the embryo transfer (from 8 am to 8 pm)
  To study when is the best moment to measure serum progesterone on the day of FET
Pregnancy outcomes after the frozen embryo transfer | from the day of the embryo transfer to 7 weeks of pregnancy
  To evaluate the on going pregnancy rate (OPR) in patients who underwent HRT FET or mNC FET. OPR is defined as a viable pregnancy at the ultrasound taken at 12 weeks of gestation that shows the presence of fetal heartbeat

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Brussels IVF, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mackens S, Santos-Ribeiro S, van de Vijver A, Racca A, Van Landuyt L, Tournaye H, Blockeel C. Frozen embryo transfer: a review on the optimal endometrial preparation and timing. Hum Reprod. 2017 Nov 1;32(11):2234-2242. doi: 10.1093/humrep/dex285. PMID 29025055
- [Background] Melo P, Chung Y, Pickering O, Price MJ, Fishel S, Khairy M, Kingsland C, Lowe P, Petsas G, Rajkhowa M, Sephton V, Tozer A, Wood S, Labarta E, Wilcox M, Devall A, Gallos I, Coomarasamy A. Serum luteal phase progesterone in women undergoing frozen embryo transfer in assisted conception: a systematic review and meta-analysis. Fertil Steril. 2021 Dec;116(6):1534-1556. doi: 10.1016/j.fertnstert.2021.07.002. Epub 2021 Aug 10. PMID 34384594
- [Background] Labarta E, Mariani G, Rodriguez-Varela C, Bosch E. Individualized luteal phase support normalizes live birth rate in women with low progesterone levels on the day of embryo transfer in artificial endometrial preparation cycles. Fertil Steril. 2022 Jan;117(1):96-103. doi: 10.1016/j.fertnstert.2021.08.040. Epub 2021 Sep 20. PMID 34548167
- [Background] Wang Z, Liu H, Song H, Li X, Jiang J, Sheng Y, Shi Y. Increased Risk of Pre-eclampsia After Frozen-Thawed Embryo Transfer in Programming Cycles. Front Med (Lausanne). 2020 Apr 8;7:104. doi: 10.3389/fmed.2020.00104. eCollection 2020. PMID 32322584
- [Background] Labarta E, Rodriguez-Varela C, Mariani G, Bosch E. Serum Progesterone Profile Across the Mid and Late Luteal Phase in Artificial Cycles Is Associated With Pregnancy Outcome. Front Endocrinol (Lausanne). 2021 Jun 10;12:665717. doi: 10.3389/fendo.2021.665717. eCollection 2021. PMID 34177806
- [Derived] Loreti S, Roelens C, Aktoz F, Niero M, De Munck N, Tournaye H, Mackens S, Blockeel C. Circadian serum progesterone variations on the day of frozen embryo transfer in a modified natural cycle protocol. Hum Reprod. 2024 May 22:deae101. doi: 10.1093/humrep/deae101. Online ahead of print. PMID 38775072